CLINICAL TRIAL: NCT02089802
Title: Optimizing Pazopanib Exposure in RCC Patients Through Therapeutic Drug Monitoring Followed by Intrapatient Dose Escalation
Brief Title: Optimizing Pazopanib Exposure in RCC Patients
Acronym: OPERA
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Early termination due to lack of recruitment
Sponsor: Interessenverband zur Qualitätssicherung der Arbeit niedergelassener Uro-Onkologen in Deutschland e. (Other)
Collaborators: OnkoDataMed GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IQUO/01 OPERA
Record Dates: First submitted 2014-03-03; First posted 2014-03-18 (Estimated); Last update posted 2017-08-18 (Actual); Status verified 2017-08

CONDITIONS: Locally Advanced Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma
Keywords: RCC
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — pazopanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Normal plasma level patients and low plasma level patients. (Experimental): 1. Patients with normal Pazopanib plasma trough levels; "normal plasma level patients" (NPLP).
  2. Patients with low Pazopanib plasma trough levels, "low plasma level patients" (LPLP).
  Interventions: Drug: Pazopanib

INTERVENTIONS:
Drug: Pazopanib

SUMMARY:
Optimization of Pazopanib Exposition in Patients with Renal Cell Carcinoma by Therapeutic Drug Monitoring followed by Individual Dose Escalation.

DETAILED DESCRIPTION:
This is an open, multi-center, intraindividual dose-optimization study. Patients with locally advanced or metastatic renal cell carcinoma receive 800 mg Pazopanib daily. After 14 days the Pazopanib plasma concentration is determined. In patients who show good tolerability and plasma trough levels of ≤ 20 µg/mLthe daily dose is increased in 200 mg steps until plasma trough levels of > 20 µg/mL are achieved or dose-limiting toxicities occur, a daily dose of 1600 mg is reached, or there is disease progression.

After each dose optimization the plasma concentration is determined after 14 days (day 11-15). If indicated, dose optimization is performed 21 days after the previous dose optimization (on day 18-24).

ELIGIBILITY:
Inclusion Criteria:

* signature of informed consent
* age ≥ 18 years
* histologically confirmed renal cell carcinoma with clear cell component and either locally progressed or metastasized
* ECOG ≤ 2
* No previous systemic therapy for locally progressed or metastasized renal cell carcinoma (previous adjuvant or neo-adjuvant therapy is permitted)
* Adequate organ function
* Female patients with child-bearing potential with negative serum pregnancy test within 2 weeks prior to first dose of study medication and adequate contraception
* Lactating females

Exclusion Criteria:

* Clinically suspected and known metastases of the central nervous system or carcinomatous meningitis except in asymptomatic patients with previously treated CNS-metastases and no necessity of steroids or anti-epileptic medication ≥ 6 months prior to start of the study medication
* Clinically significant gastrointestinal conditions with risk of increase of gastrointestinal bleeding due to (but not limited to)
* active peptic ulceration
* known intraluminal metastases with risk of bleeding
* chronic-inflammatory intestinal disease (like Morbus Crohn, ulcerative colitis) or another gastrointestinal disease with increased risk of perforation
* abdominal fistulas in anamnesis
* Clinically significant gastrointestinal conditions which can influence absorption of the IMP, among others (but not limited to)
* malabsorption syndrome
* resection of stomach or small bowel
* Current uncontrolled infection
* QTc corrected for heart frequency according to the Bazett formula
* One or more of the following cardiovascular diseases within the last 6 months in the anamnesis:
* cardiac angioplasty or coronary stent implantation
* myocardial infarction
* instable angina pectoris
* coronary-arterial bypass surgery
* symptomatic peripheral arterial occlusive disease
* Heart failure NYHA III or IV
* Poorly controlled high blood pressure
* Cerebrovascular disease, including transitory ischemic attacks, pulmonary artery embolism or untreated deep vein thrombosis within 6 months of study inclusion
* Previous major surgery or traumas within 28 days prior to start if study treatment or non-healing wound, fracture or ulcer
* Clinical signs of active bleeding or bleeding diathesis
* Known endobronchial lesions or lesions infiltrating the large lung arteries
* Haemoptyses of > 2.5 mL within 8 weeks prior to first intake of study medication
* Any other severe and/or instable medical or psychiatric pre-existing or other condition influencing patient safety, consent capacity or compliance within the study
* Incapacity or rejection to stop not allowed medication prior to first intake of study drug and pause for the duration of the trial
* Treatment with one of the following anti-tumour therapies:
* Radiation or tumour embolism within 14 days before first intake of study drug
* Chemotherapy, Immunotherapy, biological therapy, study medication or hormonal therapy within 14 days or 5 half-lives of the respective substance (whichever is longer) before first intake of the study drug. Neo-adjuvant or adjuvant therapy must have been completed for at least 6 months.
* Any present toxicity > CTC 1° from prior anti-tumour therapy and/or toxicities worsening in severity except alopecia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2014-02-25 (Actual); Primary Completion 2016-03-22 (Actual); Study Completion 2016-03-22 (Actual)

PRIMARY OUTCOMES:
Determine if in patients with a Pazopanib plasma trough level of ≤ 20 μg/mL a plasma trough level of > 20 ≤g/mL can be achieved by dose escalation. | 14 days after each dose optimization.

SECONDARY OUTCOMES:
Comparison of tumor response of patients with normal and low Pazopanib plasma trough levels. | Up to 28 days after last dose.
  Comparison of patients with normal Pazopanib plasma trough levels ("normal plasma level patients; NPLP) with patients with low Pazopanib plasma trough levels ("Low plasma level patients"; LPLP) with regard to the therapeutic result.
Objective remission rate. | Up to 28 days after last dose.
Progression free survival. | Up to 28 days after last dose.
Overall survival. | Up to 28 days after last dose.
Comparison of LPLP in whom the plasma trough level could be optimized successfully and LPLP in whom the plasma trough level could not be optimized with regard to above parameters. | Up to 28 days after last dose.
Correlation of plasma trough levels and side effects, especially high blood pressure. | Up to 28 days after last dose.
Correlation of the occurrence of high blood pressure with oncological result (response rate). | Up to 28 days after last dose.
Recording of demographic data, compliance, concomitant medication, and correlation with plasma trough levels (LPLP / NPLP). | Up to 28 days after last dose.
Examination of life quality. | Up to 28 days after last dose.

CONTACTS AND LOCATIONS:
Overall Officials: Goetz Geiges, MD, Principal Investigator — IQUO
Locations (3):
- Germany (3):
  - Gesundheitszentrum Holzminden, Holzminden, Lower Saxony
  - Private Practice Kamann, Leipzig, Saxony
  - Private Practice Geiges, Berlin